CLINICAL TRIAL: NCT04663490
Title: Neutrophil to Lymphocyte Ratio as a Predictor of Complicated Acute Diverticulitis: A Retrospective Cohort Study
Brief Title: Neutrophil to Lymphocyte Ratio as a Predictor of Complicated Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba (Other)
Responsible Party: Principal Investigator, Palacios Huatuco, General Surgeon, Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba
Other Study IDs: 0717040
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Acute Diverticulitis
Keywords: neutrophil-to-lymphocyte ratio; C-reactive protein; biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- simple acute diverticulitis: Ninety-one percent (n=295) were categorized as simple acute diverticulitis
  Interventions: Diagnostic Test: Neutrophil to Lymphocyte Ratio
- complicated acute diverticulitis: 9% (n=30) presented were categorized as complicated acute diverticulitis
  Interventions: Diagnostic Test: Neutrophil to Lymphocyte Ratio

INTERVENTIONS:
Diagnostic Test: Neutrophil to Lymphocyte Ratio — Zahorec et al. identified the neutrophil-lymphocyte ratio (NLR) as an inflammation marker in critical patients, defining as the absolute neutrophil count divided by the absolute lymphocyte count

SUMMARY:
Introduction: Various biomarkers have been studied to predict the severity of acute diverticulitis (AD), such as the leukocyte count and CRP, which are useful but lack sufficient sensitivity. The neutrophil-lymphocyte ratio (NLR) has been identified as a new inflammatory biomarker in several abdominal pathologies. However, few studies determine its association with the severity of AD. The objective of the present study was to determine the utility and diagnostic precision of NLR in complicated acute diverticulitis (cAD).

Material and methods: Descriptive, retrospective and analytical study. Patients older than 18 years with a diagnosis of AD were included, from 2013 - 2018. Demographic variables, days of hospitalization, leukocyte count, neutrophils, lymphocytes, ESR, CRP, and NLR were analyzed. The sensitivity and specificity for the diagnosis of cAD were determined using ROC curves.

DETAILED DESCRIPTION:
Introduction Acute diverticulitis (AD) is present in 10-25% of patients with diverticular disease, being most common in sigmoid colon, with around 200.000 hospitalizations yearly . As much as one fifth of patients are younger than 50 at the moment of diagnosis and around 5% under the age of 40 .

Confirming the diagnosis requires the utilization of imaging studies, therefore, American Society of Colon and Rectal Surgeons (ASCRS) established that computed tomography (CT) is the standard method for the diagnosis of AD, with a sensitivity of 98% and a specificity of 99%. The tomographic findings vary according the severity of diverticular disease, which is categorized through a modified Hinchey classification system. Approximately 10-15% of AD patients may develop complications that imply the onset of abscesses, fistulas, stenosis, obstruction and/or perforation.

Recently, interest has been raised in the role of biomarkers in diverticular disease as non-invasive, reliable, inexpensive tools that may help in the early diagnosis of complicated AD, such as C-reactive protein (CRP), useful marker in the prediction of the level of inflammation and severity of AD.

In 2001 identified the neutrophil-lymphocyte ratio (NLR) as an inflammation marker in critical patients, defining as the absolute neutrophil count divided by the absolute lymphocyte count. Over the last decade, NLR effectiveness has been recognized in various pathologies, both benign and malignant; finding that the levels of neutrophils rise as a part of the inflammatory cascade, whereas lymphocytes diminish during sepsis, making a novel subclinical biomarker with a prognostic value in oncological, cardiovascular and infectious diseases, among others. The NLR may be obtained from the blood count data, which represents a lower cost regarding other known biomarkers. It was also demonstrated that high values of NLR are associated with severe abdominal infections and worse outcomes, reason why it started to be applied as a predictor to evaluate results in surgical patients.

Currently, the debate on usefulness of NLR as a predictor of complications in AD remains open, specially, the relation to the severity of the disease, the clinical impact and the necessity of minimally invasive or emergency surgical procedures.

On the other hand, its diagnostic efficacy has not been studied even in our field. Up until now, there are only four studies published in Ireland, Israel, and South Korea. The purpose of the study was to determine the usefulness and diagnostic accuracy of NLR in complicated acute diverticulitis (cAD).

Material and methods Study population A descriptive, retrospective cohort and analytical study was undertaken. Medical histories and an electronic database from General Surgery Service were reviewed. All the patients over the age of 18 with AD diagnosis through CT were included, since January 2013 until January 2018 in a University Hospital of Cordoba, Argentina, with third level reference.

Patients were excluded if they had chronic diseases, susceptible to modify the immune inflammatory response, extra-abdominal infections, immunosuppression and neoplasias, and those who supplied incomplete data in their electronic clinical histories.

Study of variables Demographic variables (sex and age), days of inpatient stay, level of severity in diverticular process (objectified by CT) were analyzed. It was recorded the value of serum leukocyte, neutrophil, and lymphocyte concentration, Erythrocyte Sedimentation Rate (ESR), CRP and NLR at the moment of consultation on call.

Variable definition NLR: It can be obtained from the blood count (the absolute neutrophil count divided by the absolute lymphocyte count) CRP: normal value under 5 mg/l. Statistical analysis The categorical variables were expressed as frequency (percentage), the continuous variables as mean value (standard deviation, SD) or median (range) according to the distribution of data; Mann Whitney test was used to compare the continuous variables, Chi-square and Fisher's tests were used to compare categorical variables among patients with simple acute diverticulitis (sAD) and cAD. A value of p<0.05 was considered as statistically significant.

ROC (Receiver Operating Characteristic) curves were used as diagnostic tests to evaluate the diagnostic accuracy of NLR as predictor of complicated AD, determining sensitivity (Se), specificity (Sp), positive predictive value (PPV) and negative predictive value (NPV). Youden index was used to find the cut-off point with the best diagnostic yield for NLR in cAD. SPSS 26 software and GraphPad 7 software were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with a diagnosis of acute diverticulitis confirmed by computed tomography.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with hematological diseases.
* Patients with extra abdominal infections.
* Patients with oncological diseases

Ages: 18 Years to 92 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 325 patients
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Demographic variables | 2013-2018
  sex and age
inpatient stay | 2013-2018
  days
level of severity in diverticular process | 2013-2018
  confirmed by computed tomography
value of C-reactive protein | 2013-2018
  normal value under 5 mg/l
value of Neutrophil to Lymphocyte Ratio | 2013-2018
  It can be obtained from the blood count (the absolute neutrophil count divided by the absolute lymphocyte count)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria Reina Fabiola, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the study, patients were assured that the raw data would remain confidential and would not be shared.

REFERENCES:
- [Background] Weizman AV, Nguyen GC. Diverticular disease: epidemiology and management. Can J Gastroenterol. 2011 Jul;25(7):385-9. doi: 10.1155/2011/795241. PMID 21876861
- [Background] Feingold D, Steele SR, Lee S, Kaiser A, Boushey R, Buie WD, Rafferty JF. Practice parameters for the treatment of sigmoid diverticulitis. Dis Colon Rectum. 2014 Mar;57(3):284-94. doi: 10.1097/DCR.0000000000000075. No abstract available. PMID 24509449
- [Background] Barat M, Dohan A, Pautrat K, Boudiaf M, Dautry R, Guerrache Y, Pocard M, Hoeffel C, Eveno C, Soyer P. Acute colonic diverticulitis: an update on clinical classification and management with MDCT correlation. Abdom Radiol (NY). 2016 Sep;41(9):1842-50. doi: 10.1007/s00261-016-0764-1. PMID 27138434
- [Background] Wasvary H, Turfah F, Kadro O, Beauregard W. Same hospitalization resection for acute diverticulitis. Am Surg. 1999 Jul;65(7):632-5; discussion 636. PMID 10399971
- [Background] Bates DDB, Fernandez MB, Ponchiardi C, von Plato M, Teich JP, Narsule C, Anderson SW, Gupta A, LeBedis CA. Surgical management in acute diverticulitis and its association with multi-detector CT, modified Hinchey classification, and clinical parameters. Abdom Radiol (NY). 2018 Aug;43(8):2060-2065. doi: 10.1007/s00261-017-1422-y. PMID 29204676
- [Background] Kaser SA, Fankhauser G, Glauser PM, Toia D, Maurer CA. Diagnostic value of inflammation markers in predicting perforation in acute sigmoid diverticulitis. World J Surg. 2010 Nov;34(11):2717-22. doi: 10.1007/s00268-010-0726-7. PMID 20645093
- [Background] Zahorec R. Ratio of neutrophil to lymphocyte counts--rapid and simple parameter of systemic inflammation and stress in critically ill. Bratisl Lek Listy. 2001;102(1):5-14. English, Slovak. PMID 11723675
- [Background] Zahorec R. Neutrophil-to-lymphocyte ratio. Sixteen-year-long history since publication of our article in Bratislava Medical Journal. Bratisl Lek Listy. 2017;118(6):321-323. doi: 10.4149/BLL_2017_062. No abstract available. PMID 28664739
- [Background] Miyamoto R, Inagawa S, Sano N, Tadano S, Adachi S, Yamamoto M. The neutrophil-to-lymphocyte ratio (NLR) predicts short-term and long-term outcomes in gastric cancer patients. Eur J Surg Oncol. 2018 May;44(5):607-612. doi: 10.1016/j.ejso.2018.02.003. Epub 2018 Feb 13. PMID 29478743
- [Background] Reynolds IS, Heaney RM, Khan W, Khan IZ, Waldron R, Barry K. The Utility of Neutrophil to Lymphocyte Ratio as a Predictor of Intervention in Acute Diverticulitis. Dig Surg. 2017;34(3):227-232. doi: 10.1159/000450836. Epub 2016 Dec 10. PMID 27941316
- [Background] Hogan J, Sehgal R, Murphy D, O'Leary P, Coffey JC. Do Inflammatory Indices Play a Role in Distinguishing between Uncomplicated and Complicated Diverticulitis? Dig Surg. 2017;34(1):7-11. doi: 10.1159/000447250. Epub 2016 Jun 24. PMID 27336407
- [Background] Zager Y, Horesh N, Dan A, Aharoni M, Khalilieh S, Cordoba M, Nevler A, Gutman M, Rosin D. Associations of novel inflammatory markers with long-term outcomes and recurrence of diverticulitis. ANZ J Surg. 2020 Oct;90(10):2041-2045. doi: 10.1111/ans.16220. Epub 2020 Aug 28. PMID 32856387
- [Background] Mari A, Khoury T, Lubany A, Safadi M, Farraj M, Farah A, Kadah A, Sbeit W, Mahamid M. Neutrophil-to-Lymphocyte and Platelet-to-Lymphocyte Ratios Are Correlated with Complicated Diverticulitis and Hinchey Classification: A Simple Tool to Assess Disease Severity in the Emergency Department. Emerg Med Int. 2019 Aug 14;2019:6321060. doi: 10.1155/2019/6321060. eCollection 2019. PMID 31485352
- [Background] Kang HS, Cha YS, Park KH, Hwang SO. Delta neutrophil index as a promising prognostic marker of emergent surgical intervention for acute diverticulitis in the emergency department. PLoS One. 2017 Nov 1;12(11):e0187629. doi: 10.1371/journal.pone.0187629. eCollection 2017. PMID 29091955
- [Background] Agha RA, Borrelli MR, Vella-Baldacchino M, Thavayogan R, Orgill DP; STROCSS Group. The STROCSS statement: Strengthening the Reporting of Cohort Studies in Surgery. Int J Surg. 2017 Oct;46:198-202. doi: 10.1016/j.ijsu.2017.08.586. Epub 2017 Sep 7. PMID 28890409
- [Background] Jeon TJ, Park JY. Clinical significance of the neutrophil-lymphocyte ratio as an early predictive marker for adverse outcomes in patients with acute pancreatitis. World J Gastroenterol. 2017 Jun 7;23(21):3883-3889. doi: 10.3748/wjg.v23.i21.3883. PMID 28638228
- [Background] Bharucha AE, Parthasarathy G, Ditah I, Fletcher JG, Ewelukwa O, Pendlimari R, Yawn BP, Melton LJ, Schleck C, Zinsmeister AR. Temporal Trends in the Incidence and Natural History of Diverticulitis: A Population-Based Study. Am J Gastroenterol. 2015 Nov;110(11):1589-96. doi: 10.1038/ajg.2015.302. Epub 2015 Sep 29. PMID 26416187